CLINICAL TRIAL: NCT02396524
Title: Hockey Fans in Training (Hockey FIT): A Pilot Pragmatic Randomized Controlled Trial of an Exercise and Healthy Living Program for Middle-aged, Overweight and Obese Men
Brief Title: Hockey Fans in Training (Hockey FIT): A Pilot Pragmatic Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Robert Petrella, Dr. Robert J. Petrella, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: pHFIT123
Record Dates: First submitted 2015-02-26; First posted 2015-03-24 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Overweight; Obesity
Keywords: Chronic Disease; Lifestyle Intervention; Health Promotion; Sport Mentorship; Men; Health Technology; Prevention; Exercise; Diet
MeSH Terms: conditions — Overweight; Obesity; Chronic Disease; Multiple Endocrine Neoplasia Type 1; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hockey FIT program (Experimental): 12-week active phase - exercise and healthy living program (1x/week; 90 minutes/session); 40-week maintenance phase (individualized approach)
  Interventions: Behavioral: Hockey FIT Program
- Usual-care wait-list control (No Intervention): No active intervention (usual care)

INTERVENTIONS:
Behavioral: Hockey FIT Program — Active phase: a) Classroom-based education on successful weight management strategies and instruction on behaviour change techniques/dietary interventions; promote peer and other forms of social support; and b) Physical activity sessions in aerobic/strength/flexibility exercises. Maintenance phase: Participants independently set new lifestyle prescriptions and goals and track their exercise, physical activity, and healthy eating with the support of a suite of free-of-charge health technology support tools
  Other Names: Hockey Fans in Training Program; Hockey Fans in Training; Hockey FIT
  Arms: Hockey FIT program

SUMMARY:
The Hockey Fans in Training (Hockey FIT) program aims to improve overweight men's physical fitness, eating habits and health-related lifestyle choices through a lifestyle modification program in collaboration with two Ontario Hockey League teams. In this pilot pragmatic randomized controlled trial, the investigators plan to explore the potential for Hockey FIT to reduce a clinically important amount of weight, increase physical activity levels, and lead to improvements in other health-related outcomes.

DETAILED DESCRIPTION:
In the United Kingdom, the Football Fans in Training (FFIT) program was developed to encourage men to lead a healthier lifestyle through a sport-related medium. FFIT is a gender-sensitized, weight loss and healthy living program developed for delivery to overweight and obese men through professional football clubs. Published results from FFIT show that the program was able to actively recruit and engage men and for the men who participated, sustained weight loss and positive lifestyle change was observed (Hunt et al., 2014).

This study will use a two-arm, pilot pragmatic randomized controlled trial (RCT) design. The investigators will conduct the study in conjunction with two Ontario Junior A Hockey Clubs. Following assessment of eligibility and baseline measurements, men will be individually randomized (1:1; stratified by club) to either the intervention group (receiving the Hockey FIT program) or to the comparison group (usual care wait-list control). The comparison group will be offered to start the Hockey FIT program after a 12-week delay. All men (both intervention and comparison groups) will receive publicly available healthy eating and physical activity materials at baseline. Measurements will be taken at baseline and 12 weeks (both groups) and again at 12 months (intervention group only).

The results of this study will be used to inform a fully-powered RCT where the primary objective will be to determine whether, compared to the usual care wait-list control group, the Hockey FIT group will lose weight (at least 5% weight loss from baseline) at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Objectively-measured body-mass index of at least 28 kg/m2
* Clear Physical Activity Readiness Questionnaire (PAR-Q) (i.e., either by answering "No" to all questions or receiving clearance from a health care provider)

Exclusion Criteria:

* Unable to comprehend letter of information and consent documentation

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Weight loss (absolute and percentage) | 12 weeks
  Measured using digital weight scale

SECONDARY OUTCOMES:
Weight loss (absolute and percentage) | 12 months (Hockey FIT group only)
  Measured using digital weight scale
Average steps per day using pedometer | 12 weeks (& 12 months - Hockey FIT group only)
  Measured over a 7-day period using pedometers
Total physical activity in MET-minutes/week using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  International Physical Activity Questionnaire - Short Version
Time spent in sedentary activity using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by the International Physical Activity Questionnaire - Short Version
Eating habits: Fatty food score using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by the modified Dietary Instrument for Nutrition Education
Eating habits: fruit and vegetable score using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by the modified Dietary Instrument for Nutrition Education
Eating habits: sugary food score using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by the modified Dietary Instrument for Nutrition Education
Eating habits: Starting the conversation summary score using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by Starting the Conversation Dietary Assessment Tool
Alcohol consumption using recall questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by a 7-day alcohol recall (number of drinks in last 7 days)
Resting systolic blood pressure | 12 weeks (& 12 months - Hockey FIT group only)
  Measured using automated blood pressure monitor
Resting diastolic blood pressure | 12 weeks (& 12 months - Hockey FIT group only)
  Measured using automated blood pressure monitor
Waist circumference | 12 weeks (& 12 months - Hockey FIT group only)
  Measured using tape measure
Body mass index using height and weight measures | 12 weeks (& 12 months - Hockey FIT group only)
  Height will be measured with a portable stadiometer; weight will be measured with a digital weight scale
Self-esteem summary score using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Summary score from Rosenberg Self Esteem Scale
Positive affect score using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by the International Positive and Negative Affect Schedule Short Form
Negative affect score using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  Measured by the International Positive and Negative Affect Schedule Short Form
Health-related quality of life: Descriptive health state using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  EQ-5D index measured by EQ-5D-3L
Health-related quality of life: VAS using questionnaire | 12 weeks (& 12 months - Hockey FIT group only)
  EQ VAS measured by EQ-5D-3L

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Petrella, MD, PhD, Principal Investigator — University of Western Ontario, Lawson Health Research Institute
Locations (2):
- Canada (2):
  - London Knights, London, Ontario
  - Sarnia Sting, Sarnia, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blunt W, Gill DP, Sibbald SL, Riggin B, Pulford RW, Scott R, Danylchuk K, Gray CM, Wyke S, Bunn C, Petrella RJ. Optimization of the Hockey Fans in Training (Hockey FIT) weight loss and healthy lifestyle program for male hockey fans. BMC Public Health. 2017 Nov 28;17(1):916. doi: 10.1186/s12889-017-4926-z. PMID 29183291
- [Derived] Gill DP, Blunt W, De Cruz A, Riggin B, Hunt K, Zou G, Sibbald S, Danylchuk K, Zwarenstein M, Gray CM, Wyke S, Bunn C, Petrella RJ. Hockey Fans in Training (Hockey FIT) pilot study protocol: a gender-sensitized weight loss and healthy lifestyle program for overweight and obese male hockey fans. BMC Public Health. 2016 Oct 19;16(1):1096. doi: 10.1186/s12889-016-3730-5. PMID 27756351